CLINICAL TRIAL: NCT02727244
Title: Is There an Association Between Pain Catastrophizing Scale Score and Postspinal Headache in Patients Underwent Cesarean Section With Spinal Anesthesia?
Brief Title: The Association Between Pain Catastrophizing Scale Score and Postspinal Headache
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mustafa Suren, Associate Professor, Tokat Gaziosmanpasa University
Other Study IDs: 16-KAEK-071
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Pain; Headache
Keywords: Pain Catastrophizing Scale
MeSH Terms: conditions — Pain; Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: urgent or elective cesarean section — a kind of surgical procedure to deliver a baby

SUMMARY:
This study is aimed to elucidate the association between Pain Catastrophizing Scale Score and Postspinal Headache in Patients Underwent Cesarean Section With Spinal Anesthesia.

DETAILED DESCRIPTION:
This study is aimed to elucidate the association between Pain Catastrophizing Scale Score and Postspinal Headache in Patients Underwent Cesarean Section With Spinal Anesthesia. Patients were asked to fill the questionnaire booklet including Pain Catastrophizing Scale, Beck Depression Inventory and Beck Anxiety Inventory before elective cesarean section in preoperative room in operating theater. In postoperative second and fourth day, patients will call by phone and be asked to have headache or any complaints. The intensity of headache will evaluate by using visual analog scale. Age, gender, and visual analog scale scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score of I, II, III
* without a history of cerebrovascular diseases
* without any presence of psychiatric diseases

Exclusion Criteria:

* severe liver, kidney and cardiovascular diseases
* peripheral arterial diseases
* a history of allergy to local anesthetics
* patients without cooperation
* not to participate in the study
* presence of neurologic or neuromuscular diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with pregnancy whose planned to undergo urgent or elective cesarean section
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
pain catastrophizing scale score | one time in one year
  numerical value obtained using pain catastrophizing scale score

SECONDARY OUTCOMES:
Beck depression inventory | one time in one year
  numerical value obtained using Beck depression inventory
beck anxiety inventory | one time in one year
  numerical value obtained using beck anxiety inventory
visual analog scale score | one time in one year
  numerical value obtained using visual analog scale score

IPD SHARING:
Plan to Share IPD: No